CLINICAL TRIAL: NCT01620554
Title: Minimum Effective Dose-Finding Study of BF2.649, in Patients With Moderate to Severe OSA, Experiencing EDS Despite Regular Use of nCPAP, and Patients Having Refused This Therapy - Randomized, Double Blind Study With BF2.649 or Placebo
Brief Title: Dose-range Finding Study of BF2.649 Effect on Patients With Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P09-16 / BF2.649; 2010-019413-25 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obstructive Sleep Apnoea; Excessive Daytime Sleepiness
Keywords: Sleep disorder; Obstructive Sleep Apnoea; Excessive Daytime Sleepiness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence; Sleep Wake Disorders | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BF2.649 5mg (Experimental)
  Interventions: Drug: BF2.649
- BF2.649 10mg (Experimental)
  Interventions: Drug: BF2.649
- BF2.649 20mg (Experimental)
  Interventions: Drug: BF2.649
- BF2.649 40mg (Experimental)
  Interventions: Drug: BF2.649
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BF2.649 — 1 capsule per week during 2 weeks
  Other Names: Pitolisant
  Arms: BF2.649 5mg
Drug: BF2.649 — 1 capsule per week during 2 weeks
  Other Names: Pitolisant
  Arms: BF2.649 10mg
Drug: BF2.649 — 1 capsule per week during 2 weeks
  Other Names: Pitolisant
  Arms: BF2.649 20mg
Drug: BF2.649 — 1 capsule per week during 2 weeks
  Other Names: Pitolisant
  Arms: BF2.649 40mg
Drug: Placebo — 1 capsule per week during 2 weeks
  Arms: Placebo

SUMMARY:
Prospective, multicenter, double-blind, phase II, randomized, dose-response study in 5 parallel groups (dose-range).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a relatively common condition and is estimated to affect 2 to 4% of middle-aged adults

The study medication BF2.649 tested here is a novel, highly potent, selective, orally active inverse agonist at the histamine H3 receptor, therefore strengthens histaminergic transmission in the brain and increases wakefulness EDS is characterized by daytime somnolence and sudden sleep episodes. This problem has several consequences, e.g., an impairment of quality of life, an interference with activities of daily living and other handicaps in the management of social and family affairs.

The primary endpoint of this study will be measured by the change in the well-validated Epworth sleepiness scale (ESS). The ESS is a simple self-administered 8-item questionnaire. The outcome is to get an impression about the level of the daytime sleepiness in several real-life situations.

In this study, each patient will be treated during 2 weeks, and randomly assigned to one the 5 arms (BF2.649 at one of the 4 possible dosages or placebo).

The patient will then attend a end-of-treatment visit, in order to assess the particularly the ESS score.

ELIGIBILITY:
Main inclusion Criteria:

* Patient with OSA (treated or not with nCPAP) and still complaining of EDS
* Epworth Sleepiness Scale score > or = to 11

Main exclusion Criteria:

* Patient suffering from chronic severe insomnia in accordance with the International Classification of Sleep Disorders, but without OSA

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale scores (ESS) | change of ESS at 2 weeks
  ESS value compared from baseline (Day 0) and End of treatment period (Day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne De Paillette, MD, Study Director — Bioprojet
Locations (1):
- CHU de Grenoble, Grenoble, France